CLINICAL TRIAL: NCT07346833
Title: Deciphering The Role of Circulating MicroRNAs To Differentiate Psychological Disorders Among Women With Chronic Toxoplasmosis
Brief Title: Role of Circulating MicroRNAs in Differentiating Psychological Disorders Among Women With Chronic Toxoplasmosis
Status: Recruiting | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Heba M. Aboelela, Assistant Professor of Medical Parasitology, Faculty of Medicine, Benha University, Egypt, Benha University
Other Study IDs: RC 10.10.2025
Record Dates: First submitted 2025-12-21; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Toxoplasmosis
MeSH Terms: conditions — Toxoplasmosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T. gondii Seropositive Group: Women with diagnosed psychiatric disorders (Schizophrenia, MDD, or Bipolar Disorder) who test positive for anti-Toxoplasma IgG antibodies, indicating chronic infection.
  Interventions: Diagnostic Test: Circulating miRNA Expression and T. gondii Serology
- T. gondii Seronegative Group: Women with the same diagnosed psychiatric disorders who test negative for anti-Toxoplasma IgG antibodies
  Interventions: Diagnostic Test: Circulating miRNA Expression and T. gondii Serology

INTERVENTIONS:
Diagnostic Test: Circulating miRNA Expression and T. gondii Serology — Serology: ELISA testing to detect anti-Toxoplasma IgG (confirming chronic infection) and IgM (excluding acute infection).
  Genetic Analysis: Quantitative Reverse-transcriptase PCR (qRT-PCR) to measure the expression levels of a predetermined panel of plasma miRNAs.
  Psychiatric Evaluation: Clinical diagnosis according to DSM-5 criteria.

SUMMARY:
Chronic Toxoplasma gondii (T. gondii) infection is a widespread condition that can negatively affect brain function and is considered a risk factor for various psychiatric conditions, including depression and schizophrenia. This prospective observational study aims to investigate the expression levels of specific circulating microRNAs (miRNAs) in women diagnosed with schizophrenia, major depressive disorder, or bipolar disorder who also have chronic toxoplasmosis. By comparing these levels to patients without the infection, the study seeks to determine if these miRNAs can serve as biological markers to help differentiate between specific psychological disorders and identify the impact of chronic toxoplasmosis on mental health.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed psychiatric diagnosis of Schizophrenia (SCZ), Major Depressive Disorder (MDD), or Bipolar Disorder (BD) according to DSM-5 criteria.
* Seronegative for T. gondii IgM (to ensure infection is not in the acute phase).
* Signed informed consent.

Exclusion Criteria:

* Psychiatric disorders other than Schizophrenia, MDD, and Bipolar Disorder.

Seropositive for T. gondii IgM (indicating acute infection).

Refusal to participate.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of adult women (aged 18 years and older) who have been clinically diagnosed with Schizophrenia, Major Depressive Disorder, or Bipolar Disorder according to DSM-5 criteria. These patients are recruited from the psychiatric departments of Benha and Tanta Universities. Within this group, the population is divided into two cohorts: those with chronic toxoplasmosis (confirmed by the presence of anti-Toxoplasma IgG antibodies) and those without the infection. To ensure a specific focus on chronic cases, the study excludes patients with acute toxoplasmosis (IgM positive) or other unrelated psychiatric conditions. No healthy volunteers are included, as the research specifically aims to differentiate biomarkers among patients already experiencing psychological disturbances.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Plasma miRNA Expression for Detecting Chronic Toxoplasmosis in Psychiatric Patients | 2-3 Months
  The Area Under the Receiver Operating Characteristic (ROC) Curve (AUC) used to determine the diagnostic performance of circulating microRNA fold-change (measured by qRT-PCR) in discriminating between patients with and without chronic T. gondii infection (confirmed by anti-Toxoplasma IgG ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Basma Salem, MD, Principal Investigator — Assistant Professor Clinical and Chemical Pathology. Faculty of Medicine, Benha University, Egypt; Dina Abd El hadi, MD, Principal Investigator — Assistant Professor Medical Parasitology. Faculty of Medicine, Benha University, Egypt
Locations (1):
- Benha faculty of Medicine, Banhā, El Qalyoubia, Egypt